CLINICAL TRIAL: NCT04763525
Title: Stress and Biomarkers of Aging: a Novel Stress Management Program With the Cognitive Restructuring Method "Pythagorean Self-Awareness Intervention" in Healthy Individuals and in Subjects With Type 2 Diabetes Mellitus.
Brief Title: Efficacy of Pythagorean Self-Awareness for Aging Biomarkers Improvement, in T2D Patients and Healthy Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: National Hellenic Research Foundation (Other); Laikο General Hospital, Athens (Other); Aghia Sophia Children's Hospital of Athens (Other); University of Thessaly (Other)
Responsible Party: Principal Investigator, Christina Darviri, Professor of Health Promotion-Prevention and Epidemiology, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5134/5-4-19
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Mellitus; Telomere Shortening
Keywords: Stress physiology; behavioural intervention; stress management; type 2 diabetes; Pythagorean Self-Awareness
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group Pythagorean Self-Awareness in patients with type 2 diabetes (Experimental): N=21 patients with type 2 diabetes
  Interventions: Behavioral: Pythagorean Self-Awareness Intervention(PSAI)
- Intervention group Pythagorean Self-Awareness for healthy individuals (Experimental): N=27 healthy individuals
  Interventions: Behavioral: Pythagorean Self-Awareness Intervention(PSAI)

INTERVENTIONS:
Behavioral: Pythagorean Self-Awareness Intervention(PSAI) — The PSAI is a mental, stress-management technique that promotes self-awareness, cognitive reconstruction and self-improvement based on the Golden Verses moral framework of the ancient Greek philosopher Pythagoras. The individual must practice the technique twice daily( at bed-time and in the morning, every day, at home) and through a 3-stage internal dialogue (recall of daily events, inspection of related thoughts and emotions and self-appraisal)is encouraged to detect wrong choices and unhealthy behaviours and initiate self-correction towards a healthier lifestyle.

SUMMARY:
The present study explored the effects of the implementation of the Pythagorean Self Awareness Intervention (PSAI) on the dynamics of stress-related aging factors of immune cells in healthy volunteers and a cohort patients with type 2 diabetes mellitus . The primary aim was to evaluate the effectiveness of PSAI on two key biomarkers of biological age, telomere length and proteasome levels, indicative of the crosstalk between cellular oxidative status and replicative potential, with respect to metabolic, hormonal and mental status changes. Secondary aims of this study included reduction of depression, perceived stress, anxiety and the establishment of lifestyle changes to enhance the quality of everyday life, including better quality of sleep, eating behaviours and an overall healthier status.

DETAILED DESCRIPTION:
Study design This non randomized non blinded parallel trial was conducted at the Laiko Hospital of Athens, Diabetes Centre, First Department of Propaedeutic Internal Medicine of Attica, Greece, from 4.10.2018 to 26.11.2019. The study protocol was approved by the Ethics Committee of the Laiko Hospital (protocol number 5134/5-4-19) and was in accordance with the declaration of Helsinki. All participants were enlisted in the study only after being fully informed by the researcher about the aims and procedures of the research and submitting written consent.

Procedures Patients eligible for the above mentioned criteria were randomized in two groups: the group of healthy adult volunteers, and adults with type 2 diabetes who attended the outpatient diabetes clinic. This study was non-blinded, as patients and researchers were aware of the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* adequate knowledge of the Greek language
* For participants with T2DM, a minimum of 3-month stable antidiabetic, hypolipidemic and antihypertensive treatment
* habitants of Athens, Greece

Exclusion Criteria:

* participation in other stress management program
* corticosteroid intake
* diagnosis of psychiatric co-morbidity or autoimmune disease
* change in antidiabetic, hypolipidemic, and antihypertensive treatment within the previous 3 months
* patients with type 2 diabetes treated with insulin

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Determination of telomeres' length | 2 months
  Extracted DNA from Peripheral blood mononuclear cells isolated from total blood
Determination of telomeres' length | 6 months
  Extracted DNA from Peripheral blood mononuclear cells isolated from total blood
Determination of 20S proteasome concentration | 6 months
  Protein extracts from Peripheral blood mononuclear cells isolated from total blood
Healthy Lifestyle and Personal Control Questionnaire | 6 months
  Self-report questionnaire for the evaluation of a healthy lifestyle with the instrument Healthy Lifestyle and Personal Control Questionnaire that explores five dimensions of lifestyle (Organized Physical Exercise, Social Support and Mental Control, Daily Routine, Dietary Harm Avoidance, Dietary Healthy Habits).Scores range from 26 to 104 with higher scores indicating a healthier lifestyle.
Glycosylated haemoglobin | 6 months
  total blood

SECONDARY OUTCOMES:
Hair cortisol concentration | 6 months
  Hair specimens from the posterior vertex of the scalp, three cm proximal to scalp
Total Body Water | 6 months
  Total Body Water will be reported in percent and it will be measured by the device TANITA BC418 (Tanita Cooperation, Tokyo, Japan),
Fat Free Mass | 6 months
  Fat Free Mass will be reported in kilograms,and it will be measured by the device TANITA BC418 (Tanita Cooperation, Tokyo, Japan),
Fat Mass | 6 months
  Fat Mass will be reported in percentage and it will be measured by the device TANITA BC418 (Tanita Cooperation, Tokyo, Japan),
Visceral fat | 6 months
  Visceral fat will be reported in cm ^2 and it will be measured by the device TANITA BC418 (Tanita Cooperation, Tokyo, Japan)
Trunk fat | 6 months
  Trunk fat will be reported in percentage and it will be measured by the device TANITA BC418 (Tanita Cooperation, Tokyo, Japan)
Body Mass Index | 6 months
  Weight and height will be combined to report BMI in kg/m^2
Depression Anxiety Stress Scale | 6 months
  Self-referential symptoms of depression, anxiety and stress with the instrument Depression-Anxiety-Stress Scale-21 Three scores(Depression, Anxiety, Stress). Depression score ranging from 0 to 42, Anxiety score ranging from 0-42, Stress score ranging from 0-42. We expect reduction.
Perceived Stress Scale | 6 months
  Evaluation with the self-referential instrument the Perceived Stress Scale. Score ranging from 0 to 56 with higher score indicating higher perceived stress. We expect reduction.
Self-referential quality of sleep | 6 months
  Evaluation of sleep quality with the instrument Greek version Pittburgh Sleep Quality Index. Score ranging from 0 to 21. Score higher than 5 indicates poor sleep quality. We expect reduction.
Self-referential Internal Health Locus of Control | 6 months
  Evaluation of internal health locus with the instrument Health Locus of Control. Score ranging from 6 to 36 with higher scores indicating higher self-control over the individual's health. We expect increase.
Self-referential External and chance Health Locus of Control | 6 months
  Evaluation of External health locus of control and chance, with the instrument Health Locus of Control. Score ranging from 6 to 36 for each dimension. Higher score means that the individual perceives that his/her health is controlled by external factors and chance.We expect reduction.
Self-referential health locus of control Powerful others | 6 months
  Evaluation of health locus of control for Powerful others with the instrument Health Locus of Control. Score ranging from 6 to 36.Higher score means that the individual perceives that his/her health is controlled by powerful others such as health personnel.We expect reduction.
Evaluation of verbal memory | 6 months
  Assessment of verbal memory with the cognitive test California Verbal Learning test. Score ranging from 0 to 90 with higher score indicating better verbal memory. We expect increase.
Evaluation of visuospatial memory | 6 months
  Assessment of visuospatial memory with the cognitive test Brief Visuospatial Memory test-Revised. Score ranging from 0 to 36 with higher score indicating better visuospatial memory.We expect increase.
Evaluation of speed processing information | 6 months
  Assessment of speed processing of information with the cognitive test Symbol Digits Modality test. Score ranging from 0 to 95 with higher score indicating higher speed processing of information.We expect increase.
Fatigue | 6 months
  Assessment of physical, mental and brain fatigue with a visual analogue scale with minimum as 0 indicating no fatigue at all and maximum 10 indicating high degree of fatigue. We expect reduction.
Perimeter of the waist | 6 months
  Perimeter will be reported in centimeters
Perimeter of the neck | 6 months
  Perimeter will be reported in centimeters
Perimeter of the hips | 6 months
  Perimeter will be reported in centimeters
Extracellular water | 6 months
  Extracellular water will be reported in percentage and with be assessed by a device of bioelectrical impedance technology by BIOTEKNA©, Biomedical Technologies, Venice, Italy
Intracellular water | 6 months
  Intracellular water will be reported in percentage and it will be measured by a device of bioelectrical impedance technology by BIOTEKNA©, Biomedical Technologies, Venice, Italy

CONTACTS AND LOCATIONS:
Overall Officials: Christina Darviri, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- General University Laiko Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
The data will be made available upon study publication.

REFERENCES:
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838
- [Background] de Magalhaes JP, Passos JF. Stress, cell senescence and organismal ageing. Mech Ageing Dev. 2018 Mar;170:2-9. doi: 10.1016/j.mad.2017.07.001. Epub 2017 Jul 5. PMID 28688962
- [Background] Weber D, Stuetz W, Toussaint O, Debacq-Chainiaux F, Dolle MET, Jansen E, Gonos ES, Franceschi C, Sikora E, Hervonen A, Breusing N, Sindlinger T, Moreno-Villanueva M, Burkle A, Grune T. Associations between Specific Redox Biomarkers and Age in a Large European Cohort: The MARK-AGE Project. Oxid Med Cell Longev. 2017;2017:1401452. doi: 10.1155/2017/1401452. Epub 2017 Jul 19. PMID 28804532
- [Background] Chondrogianni N, Stratford FL, Trougakos IP, Friguet B, Rivett AJ, Gonos ES. Central role of the proteasome in senescence and survival of human fibroblasts: induction of a senescence-like phenotype upon its inhibition and resistance to stress upon its activation. J Biol Chem. 2003 Jul 25;278(30):28026-37. doi: 10.1074/jbc.M301048200. Epub 2003 May 7. PMID 12736271
- [Background] Puhlmann LMC, Valk SL, Engert V, Bernhardt BC, Lin J, Epel ES, Vrticka P, Singer T. Association of Short-term Change in Leukocyte Telomere Length With Cortical Thickness and Outcomes of Mental Training Among Healthy Adults: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e199687. doi: 10.1001/jamanetworkopen.2019.9687. PMID 31553468
- [Background] Diaz-Ruiz A, Guzman-Ruiz R, Moreno NR, Garcia-Rios A, Delgado-Casado N, Membrives A, Tunez I, El Bekay R, Fernandez-Real JM, Tovar S, Dieguez C, Tinahones FJ, Vazquez-Martinez R, Lopez-Miranda J, Malagon MM. Proteasome Dysfunction Associated to Oxidative Stress and Proteotoxicity in Adipocytes Compromises Insulin Sensitivity in Human Obesity. Antioxid Redox Signal. 2015 Sep 1;23(7):597-612. doi: 10.1089/ars.2014.5939. Epub 2015 Mar 31. PMID 25714483
- [Background] Tsoli S, Vasdekis S, Tigani X, Artemiadis A, Chrousos G, Darviri C. A novel cognitive behavioral treatment for patients with chronic insomnia: A pilot experimental study. Complement Ther Med. 2018 Apr;37:61-63. doi: 10.1016/j.ctim.2018.01.015. Epub 2018 Feb 1. PMID 29609939
- [Background] Charalampopoulou M, Bacopoulou F, Syrigos KN, Filopoulos E, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on breast cancer patients undergoing adjuvant therapy: A pilot randomized controlled trial. Breast. 2020 Feb;49:210-218. doi: 10.1016/j.breast.2019.12.012. Epub 2019 Dec 20. PMID 31901782
- [Background] Darviri C, Alexopoulos EC, Artemiadis AK, Tigani X, Kraniotou C, Darvyri P, Chrousos GP. The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ): a novel tool for assessing self-empowerment through a constellation of daily activities. BMC Public Health. 2014 Sep 24;14:995. doi: 10.1186/1471-2458-14-995. PMID 25253039